CLINICAL TRIAL: NCT05249673
Title: Effects of Global Postural Reeducation Versus Neck Stabilization Training on Text Neck Syndrome
Brief Title: Global Postural Reeducation Versus Neck Stabilization Training on Text Neck Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AH/21/0131/SanaMubarak
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Neck Syndrome
Keywords: Text neck syndrome, REBA questionnaire, Turtle neck posture.

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- global postural reeducation (Experimental): global postural reeducation (GPR) interventions will last 9 sessions, 1 hour each, with one-to-one supervision, once or twice a week according to the participant's needs. All participants will receive advice to follow written ergonomic suggestions and to repeat the exercises in the first physical therapy session at home twice a week for 15 minutes. Each group will get a home exercise program, which will differ according to the type of treatment received. Participants in the GPR group will execute one "posture" routine.
  Interventions: Other: global postural reeducation
- neck stabilization training (Active Comparator): Each exercise session will be comprised of 10-minute warm-up exercises, 40-minute stabilization exercises, and 10-minute cool-down and stretching exercises, including neck and shoulder girdle muscles. The whole program will be carried out 3 days per week for 4 weeks.The participants will be asked to maintain the positions and contractions during the exercises and throughout the day as much as possible. The combination and progression of the exercises will be designed according to condition of the patient.
  Interventions: Other: neck stabilization training

INTERVENTIONS:
Other: global postural reeducation — GPR interventions will last 9 sessions, 1 hour each, with one-to-one supervision, once or twice a week according to the participant's needs. All participants will receive advice to follow written ergonomic suggestions and to repeat the exercises in the first physical therapy session at home twice a week for 15 minutes. Each group will get a home exercise program, which will differ according to the type of treatment received. Participants in the GPR group will execute one "posture" routine.
  Other Names: posture training
  Arms: global postural reeducation
Other: neck stabilization training — Each exercise session will be comprised 10-minute warm-up exercises, 40-minute stabilization exercises, and 10-minute cool-down and stretching exercises, including neck and shoulder girdle muscles. The whole program will be carried out 3 days per week for 4 weeks.
  performed. The participants will be asked to maintain the positions and contractions during the exercises and throughout the day as much as possible. The combination and progression of the exercises will be designed according to condition of the patient.
  Arms: neck stabilization training

SUMMARY:
The study will be randomized control trial. The study will be conducted in Iqbal Mehmooda Trust Hospital. Group A will be treated with global postural reeducation. Group B will be treated with neck stabilization training. Non probability consecutive sampling technique will be used. Patient below 20-40 years, participants who use smart phones for 8 hours per day(guidelines), angle of forward head pasture above 15, screening picture tool.

Neurological defects, trauma, tumor, shoulder injury, cervical disc disease. REBA questionnaire, NDI, Goniometry, NPRS will be used as a tool. The global postural reeducation will be applied on group A while neck stabilization training will be applied on group B. The aim of this study will be to compare the effects of of global postural reeducation and neck stabilization training on text neck syndrome.

DETAILED DESCRIPTION:
''Text neck syndrome'' describes the neck pain and looking down at the smart gadgets repeatedly and for prolonged duration that leads to damage of various structures. The cervical spine consists of bundles of nerves, bones, joints and muscles. If nerves are compressed then pain can radiate to shoulder, arm and hand. 79% of the population between the age of 18-44 use their cell phones almost all the time except only 2 hours of their walking time without the usage of their cell phones. The forward head posture/Turtle neck posture causes strain on the muscles, ligaments and joints that leads to compression of nerves and it causes tingling and numbness in the hands. The usage of smart gadgets for prolonged duration has negative impact on our anxiety and depression. Excessive use of smart phones leads to postural problems like forward neck posture, slouched posture or rounded shoulders.

ELIGIBILITY:
Inclusion Criteria:

* Patient below 20-40 years
* Participants who use smart phones for 8 hours per day(guidelines)
* Angle of forward head posture above 15
* Screening picture tool

Exclusion Criteria:

* Neurological defects
* Trauma
* Tumor
* Shoulder injury
* Cervical disc disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
REBA questionnaire to measure body position on work station. | 6 weeks
  The Rapid Entire Body Assessment (REBA) was developed to "rapidly" evaluate the risk of musculoskeletal disorders (MSD) associated with certain job tasks. The change will be assessed from Baseline and end of treatment.
neck disability index to measure function of neck. | 6 weeks
  NDI questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. It had 10 sections with total 50 scores. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. 0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation. The change will be assessed from Baseline and end of treatment.
Numeric pain rating scale to measure pain. | 6 weeks
  this scale is used for pain. Scale consists of 4 questions regarding actual pain level, zero indicates no pain and 10 indicates worst pain imaginable. The change will be assessed from Baseline and end of treatment.

SECONDARY OUTCOMES:
Neck Ranges (Flexion, Extension, Rotation and Side bending) | 6 weeks
  Goniometer is used to measure the ranges of neck region (neck flexion, extension, rotation and side bending). The change will be assessed from Baseline and end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal investigator
Locations (1):
- Sana Mubarak, Lahore, Lahore,Punjab,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No